CLINICAL TRIAL: NCT00037700
Title: Evaluation of the Efficacy of Combination Treatment With Anakinra and Pegsunercept in Improving Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Organization: Swedish Orphan Biovitrum (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20000198
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Interleukin 1 Receptor Antagonist Protein; PEGylated soluble tumor necrosis factor receptor I

INTERVENTIONS:
Drug: anakinra
Drug: pegsunercept

SUMMARY:
The purpose of this study is to evaluate the effect of anakinra (IL-1 ra) and pegsunercept (PEG sTNF-RI) when they are used together in improving the signs and symptoms of rheumatoid arthritis. The study will also evaluate the safety of the combination treatment and its effect on slowing down bone and joint destruction due to rheumatoid arthritis. The results will be compared to the effect when only 1 single medication (anakinra or pegsunercept) is used.

ELIGIBILITY:
* diagnosed with rheumatoid arthritis for at least 6 months
* must be taking methotrexate * must not take DMARDS other than methotrexate during the study
* must not have had previous treatment with and protein-based TNF-alpha inhibitor (eg. etanercept, infliximab, PEG sTNF-RI, or D2E7)
* must not have had previous treatment with anakinra
* subjects must meet tender and swollen joint requirements at screening, have morning stiffness, and/or have elevated acute phase reactants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com